CLINICAL TRIAL: NCT02544126
Title: Computer-Based Intervention in HIV-Positive Young Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Melissa Pinto, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00080145
Record Dates: First submitted 2015-09-04; First posted 2015-09-09 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: HIV; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- eSMART-MH (Experimental): HIV+ young adults will be randomized to receive Electronic Self-Management Resource Training for Mental Health (eSMART-MH)
  Interventions: Device: Electronic Self-Management Resource Training for Mental Health
- Attention Control (Active Comparator): HIV+ young adults will be randomized to receive screen-based health education
  Interventions: Behavioral: Screen-based health education

INTERVENTIONS:
Device: Electronic Self-Management Resource Training for Mental Health — eSMART-MH is a software, which is set in a 3-D virtual primary care office environment in which a subject interacts with avatar virtual healthcare staff (medical receptionist, medical assistant, providers, and a virtual healthcare coach). The avatars are programed to behave like humans. The subject moves through the 3-D virtual primary care office and encounters virtual healthcare staff and providers. The subject practices discussing depressive symptoms with avatar healthcare providers and practices self-management skills related to symptoms of depression.The subject also interacts with the health care coach. The health care coach provides the subject with real-time strategies to enhance communication with healthcare providers during their virtual office visit. Overtime, coaching is decreased to build the the subject's self-confidence. eSMART-MH will be used once a month, for three months.
  Other Names: eSMART-MH
  Arms: eSMART-MH
Behavioral: Screen-based health education — Screen-based health education will be used and cover topics like depression, nutrition, physical activity, and sleep hygiene at the same frequency as the eSMART-MH intervention, which is used once a month, for three months.
  Arms: Attention Control

SUMMARY:
The purpose of this study is to investigate how working with a computer program may affect mood, feelings, overall health, and markers in blood in young adults with HIV.

DETAILED DESCRIPTION:
Depression frequently occurs in young adults with HIV infection. When young adults with HIV experience depression, they are less likely to take their prescribed antiretroviral therapy (ART). When HIV occurs simultaneously with depression, individuals are more likely to have indicators in their blood that are linked risk for developing other illnesses in the future. The purpose of this project is to examine the ability of an avatar-based intervention, called eSMART-MH, to decrease depressive symptoms in HIV-positive depressed young adults.

ELIGIBILITY:
Inclusion Criteria:

* 23-53 years of age
* Fluent in English
* Be able to view images and text on a computer screen and hear audio using a headset
* Have a diagnosis of unipolar depression or have significant depressive symptoms noted in the electronic medical record (EMR) or referred to the study by a provider at the Grady Ponce de Leon Clinic because of their depressive symptoms
* Receive care at Ponce de Leon Center and at least 1 scheduled HIV medical appointment in the last 6 months
* Reside in the Atlanta, Georgia area
* Have a valid telephone number and email address
* Answer all items correctly on consent post-test

Exclusion Criteria:

* Diagnosis of bipolar depression
* Deaf, blind or unable to understand spoken English
* Currently pregnant, history of pregnancy within the last year or plan to become pregnant within the next 4 months
* Plan to move from the Atlanta, Georgia area within four months of study enrollment
* Taking corticosteroids or disease-modifying anti-rheumatic drugs
* If on antidepressant medication, taking it for less than 1 month
* Fail to pass post-consent test after three attempt

Ages: 23 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in the Patient Health Questionnaire (PHQ-9) | Baseline, 3 months
  The PHQ-9 is a 9-item self-report measure of depressive symptoms which asks participants to rate the frequency of depression symptoms over the past 2 weeks from 0 (not at all) to 3 (nearly every day). Scores range from 0 to 27, with higher scores reflecting greater severity of depressive symptoms.
Change in the General Well-Being Schedule (GWS) | Baseline, 3 months
  The GWS is an 18-item self-report measure that examines the subjective feelings of psychological well-being and distress which asks participants to rate each question in relationship to their feelings over the past 4 weeks on a 6-grade Likert scale. The last four items ask respondents to supply ratings on a 1-10 scale. Score range will be transformed into a the scale score on a continuum from 0 to 100, with higher scores reflecting a better well being of the participant.
Change in Center for Disease Control Health Related Quality of Life-4 (CDC HRQOL-4) | Baseline, 3 months
  CDC HRQOL-4 is self-report measures quality of life over the last 30 days in the domains of physical and mental health and asks participants 4 core questions including one health status measure (self-rated health) and three HRQOL measures (recent physical health, recent mental health, and recent activity limitation). The scoring used is with a summary "unhealthy days" index, computed by adding a respondent's physically and mentally unhealthy days, with a maximum of 30 for one person.
Change in the Quality of Life Enjoyment Scale (Q-LES-Q-SF) | Baseline, 3 months
  Q-LES-Q-SF is a 16 item self-report measure that assesses the quality of life satisfaction in multiple domains of functioning which asks participants to rate how satisfied they have been with various aspects of their life over the last week, rating on a 1-5 Likert-type scale. Scores range from 16 to 80, with higher scores reflecting less enjoyment and satisfaction.

SECONDARY OUTCOMES:
Medication Adherence | Baseline, 3 months
  Pill counts for antiretroviral therapy (ART) and medication for mood (if ordered) will be measured through examining pills consumed compared to the doses prescribed.
Change in plasma interleukin-6 (IL-6) levels | Baseline, 3 months
  IL-6 is circulating inflammatory biomarker. The plasma concentrations of IL-6 will be assessed using commercial enzyme-linked immunoassay (ELISA) kits.
Change in cluster of differentiation 4 (CD4) Count | Baseline, 3 months
  CD4 is a glycoprotein found on the surface of immune cells such as T helper cells, monocytes, macrophages, and dendritic cells and is a measure for how well the immune system is working. CD4 T-cell will be assessed using flow cytometry and healthy adult/adolescent ranges from 500 cells/mm^3 to 1,200 cells/mm^3.
Change in Log HIV Viral Load | Baseline, 3 months
  Viral load measures the amount of HIV's genetic material in a blood sample. The results of a viral load test are described as the number of copies of HIV RNA in a milliliter of blood. For example, a viral load of 10,000 would be considered low; 100,000 would be considered high. Viral load changes can be very large, so they are sometimes quantified using the powers of ten, or 'log scale'. A 1-log change is the same as a ten-fold change (so 5000 to 50,000 or vice versa).
Change of plasma brain-derived neurotrophic factor (BDNF) levels | Baseline, 3 months
  BDNF is a protein that acts on certain neurons of the central nervous system and the peripheral nervous system, helping to support the survival of existing neurons, and encourage the growth and differentiation of new neurons and synapses. The plasma concentrations of BDNF will be assessed using commercial enzyme-linked immunoassay (ELISA) kits.
Change in Fibrinogen levels | Baseline, 3 months
  Fibrinogen is a hepatic-derived factor directly involved in clotting and in the viscosity characteristics of blood flow. It binds to platelets and contributes to their aggregation, promotes fibrin formation and is also an acute phase reactant that is increased in inflammatory states. The plasma concentrations of fibrinogen antigen will be assessed using the immunochemistry.
Change in plasma oxytocin levels | Baseline, 3 months
  Oxytocin, a chemical composed of a chain of amino acids, is a substance that has multiple physiological functions within the human body. These functions include roles as both a hormone as well as a neurotransmitter. The plasma concentrations of oxytocin will be assessed using commercial enzyme-linked immunoassay (ELISA) kits.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa D Pinto, PhD,RN,FAAN, Principal Investigator — Emory University